CLINICAL TRIAL: NCT02481362
Title: Food Choices in Healthy Weight Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UTK IRB-15-02330-XP
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Addictive Behavior; Food Preferences; Food Habits; Healthy; Habituation
MeSH Terms: conditions — Behavior, Addictive; Food Preferences; Feeding Behavior; Substance-Related Disorders | interventions — Prunus armeniaca extract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Order 1 (Active Comparator): Order for sessions: Cake, apricots
  Interventions: Other: CAKE; Other: APRICOTS
- Order 2 (Active Comparator): Order for sessions: apricots, Cake
  Interventions: Other: CAKE; Other: APRICOTS

INTERVENTIONS:
Other: CAKE — For the CAKE condition, participants will play a computer task to earn points for cake that they can consume.
Other: APRICOTS — For the APRICOTS condition, participants will play a computer task to earn points for apricots that they can consume.

SUMMARY:
This study will examine differences in habituation to foods high in sugar and fat content versus those that are not, in normal weight women.

DETAILED DESCRIPTION:
Participants will complete two experimental sessions, in which habituation to chocolate cake and dried apricots will be measured, with each session measuring habituation rate to one food. Upon arrival to the session, participants will write down what they have consumed and the minutes of physical activity they have engaged in during the previous 24 hours. Participants will rate their feelings of hunger and fullness using a 100mm VAS. They will also rank their liking of the food being used in the session using a 100mm VAS. Participants will be given a peanut butter flavored granola bar, containing 190 kcal, and be instructed to consume all of the bar.

Next, participants will complete a computer generated task to measure habituation to a food (chocolate cake or apricots). The computer task will be programmed at a variable interval of 120 ± 42 seconds (VI-120) reinforcement schedule, so that participants will be rewarded one point for the first response made after approximately 120s have passed. The computer task consists of two squares, one that flashes red every time a mouse button is pressed and another square that flashes green when a point is earned. The habituation phase will be 24 minutes, divided into 12, 2-minute trials, during which participants can earn points towards access to 75 kcal portions of the food that is being measured. Participants will receive the food immediately after each point is earned to consume and can continue to play the computer task while eating. Participants will be instructed that when they no longer want to earn access to the food they can go to another table and engage in the activities provided (i.e., reading magazines). After the computer task, participants will rate their feeling of hunger, fullness, and liking of the food. During the computer task the number of consecutive two-minute time blocks before responding ceases, as well as the overall pattern of responding, will be measured.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) 18.5 to 24.9 kg/m2
* nonsmokers
* not allergic to the foods used in the investigation
* must like the foods in the investigation (scoring > 50 mm on a visual analogue scale [VAS])
* be willing to consume the foods
* not have dietary restrictions
* not be a restrained eater (scoring > 12 on the Three Factor Eating Scale)
* not be on medications that influence appetite
* not planning to change their diet or physical activity during the time frame of their study participation
* not dieting or trying to lose weight.

Exclusion Criteria:

* BMI outside of the range 18.5-24.9
* smoker
* food allergies
* does not like the foods used in the study
* has dietary restrictions
* is a restrained eater
* on medications that may influence appetite
* planning on changing diet or physical activity during time frame of the study
* dieting
* trying to lose weight

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Grams of consumption of cake | 60 minutes
  Amount of cake consumed will be measured using the following formula: amount of cake before consumption (first weight) - amount of cake following consumption (second weight).
Grams of consumption of apricots | 60 minutes
  Amount of apricots consumed will be measured using the following formula: amount of apricots before consumption (first weight) - amount of apricots following consumption (second weight).

CONTACTS AND LOCATIONS:
Overall Officials: Hollie Raynor, PhD, Principal Investigator — University of Tennessee, Knoxville
Locations (1):
- Healthy Eating and Activity Laboratory, University of Tennessee, Knoxville, Tennessee, United States

REFERENCES:
- [Background] Epstein LH, Temple JL, Roemmich JN, Bouton ME. Habituation as a determinant of human food intake. Psychol Rev. 2009 Apr;116(2):384-407. doi: 10.1037/a0015074. PMID 19348547
- [Background] Epstein LH, Carr KA, Cavanaugh MD, Paluch RA, Bouton ME. Long-term habituation to food in obese and nonobese women. Am J Clin Nutr. 2011 Aug;94(2):371-6. doi: 10.3945/ajcn.110.009035. Epub 2011 May 18. PMID 21593492
- [Background] Goldfield GS, Legg C. Dietary restraint, anxiety, and the relative reinforcing value of snack food in non-obese women. Eat Behav. 2006 Nov;7(4):323-32. doi: 10.1016/j.eatbeh.2005.11.006. Epub 2005 Nov 28. PMID 17056408
- [Background] Franko DL, Wolfe BE, Jimerson DC. Elevated sweet taste pleasantness ratings in bulimia nervosa. Physiol Behav. 1994 Nov;56(5):969-73. doi: 10.1016/0031-9384(94)90331-x. PMID 7824599
- [Background] Deglaire A, Mejean C, Castetbon K, Kesse-Guyot E, Hercberg S, Schlich P. Associations between weight status and liking scores for sweet, salt and fat according to the gender in adults (The Nutrinet-Sante study). Eur J Clin Nutr. 2015 Jan;69(1):40-6. doi: 10.1038/ejcn.2014.139. Epub 2014 Jul 30. PMID 25074389
- [Background] McGloin AF, Livingstone MB, Greene LC, Webb SE, Gibson JM, Jebb SA, Cole TJ, Coward WA, Wright A, Prentice AM. Energy and fat intake in obese and lean children at varying risk of obesity. Int J Obes Relat Metab Disord. 2002 Feb;26(2):200-7. doi: 10.1038/sj.ijo.0801883. PMID 11850751
- [Background] Gearhardt AN, Roberto CA, Seamans MJ, Corbin WR, Brownell KD. Preliminary validation of the Yale Food Addiction Scale for children. Eat Behav. 2013 Dec;14(4):508-12. doi: 10.1016/j.eatbeh.2013.07.002. Epub 2013 Jul 21. PMID 24183146
- [Background] Gearhardt AN, White MA, Masheb RM, Morgan PT, Crosby RD, Grilo CM. An examination of the food addiction construct in obese patients with binge eating disorder. Int J Eat Disord. 2012 Jul;45(5):657-63. doi: 10.1002/eat.20957. Epub 2011 Aug 30. PMID 22684991
- [Background] Ridgway PS, Jeffrey DB. A comparison of the Three-Factor Eating Questionnaire and the Restraint Scale and consideration of Lowe's Three-Factor Model. Addict Behav. 1998 Jan-Feb;23(1):115-8. doi: 10.1016/s0306-4603(97)00031-2. PMID 9468749